CLINICAL TRIAL: NCT02803489
Title: Evaluation of the Performance of an e-Health System Comprising Tele-monitoring / Tele-notification and Tele-coaching in Ambulatory Multi-morbid Adult Patients
Brief Title: Evaluation of the Performance of an e-Health System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion rate too low & investigators enable to recruit new patients rapidly
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Inferential (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALMED-14-MD-051
Record Dates: First submitted 2016-05-23; First posted 2016-06-17 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Diseases
Keywords: chronic heart failure; chronic obstructive pulmonary disease; diabetes
MeSH Terms: conditions — Chronic Disease; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- medical device intervention (Experimental)
  Interventions: Device: medical device intervention

INTERVENTIONS:
Device: medical device intervention
  Other Names: Nomhad Mobile - Nomhad Chronic

SUMMARY:
Prospective, non-randomized, open-label, pilot study conducted in a single group of 30 evaluable patients, i.e. patients completing an approximate 3 month follow-up.

DETAILED DESCRIPTION:
The eHealth system developed in the present study is dedicated to multimorbid patients' follow-up. The medical device consists in Telemonitoring, Telenotification and Telecoaching. It aims to both increase patient autonomy, with regard to management of his/her pathologies, and facilitate coordination between health professionals.

By providing patients with tools enabling early detection of clinical worsening combined with an appropriate management, the medium and long-term objectives are to reduce hospitalizations and improve health status and quality of life of these patients at home.

In the first instance, the only objective of the present study is to evaluate the performance and feasibility of implementation of the device. This evaluation is based on a comparison between the telenotifications generated by the software and those calculated from the raw data captured by the software.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting all the following characteristics are eligible for inclusion:

1. Adult (>18 yrs), male or female
2. Presenting at least two chronic diseases among the following three: chronic heart failure (CHF), chronic obstructive pulmonary disease (COPD), diabetes
3. Having been hospitalized in the CHANGE or in any other medical care center (hospital or private clinic) for acute decompensation of CHF or exacerbation of COPD at least once during the 12 months prior to inclusion
4. Able to speak and understand French to a satisfactory standard
5. Having a phone land line
6. Capable of understanding and accepting the study constraints
7. Having signed a written informed consent after a full explanation of the study by the investigator prior to inclusion

Exclusion Criteria:

Patients presenting any one of the following characteristics are not eligible for inclusion:

1. Pregnant or breast-feeding woman
2. Institutionalized
3. Having a life expectancy of less than 3 months
4. Receiving or having received chemotherapy or radiotherapy for cancer within the past 6 months
5. Undergoing dialysis for chronic renal insufficiency
6. Presenting a condition likely to hamper accomplishment of the study procedures, such as chronic alcoholism, drug or solvent addiction, uncontrolled psychiatric disease or severe cognitive deficiency
7. Not covered by French Social Security
8. Participating or having participated in another interventional trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the tele-notifications | through study completion, an average of 11 months

SECONDARY OUTCOMES:
Sensitivity and specificity of the STABILITY SYSTEM INDICATORS | through study completion, an average of 11 months
Specific self-administered questionnaires about Ease of Use/Usefulness/Satisfaction for each category of user | through study completion, an average of 11 months
Acceptability of the system by patients regarding transmission of measured parameters | through study completion, an average of 11 months
  Mean number of transmission of measured parameters: real versus theoretical.
Acceptability of the system by patients: mean number of participation in virtual classroom session | through study completion, an average of 11 months
Acceptability of the system by patients: mean duration of participation in virtual classroom session | through study completion, an average of 11 months
Acceptability of the system by patients: mean number of consultations of modules providing medical information | through study completion, an average of 11 months
Acceptability of the system by patients: cumulative time spent on consultations of modules providing medical information | through study completion, an average of 11 months
Acceptability of the system by patients: mean duration of phone contacts by type (planned, for notification management, incoming) | through study completion, an average of 11 months
Acceptability of the system by patients: mean number of phone contacts by type (planned, for notification management, incoming) | through study completion, an average of 11 months
Acceptability of the system by patients: comparison of real planned phone contacts versus theoretical | through study completion, an average of 11 months
Acceptability of the system by physicians: mean number of connections | through study completion, an average of 11 months
Acceptability of the system by physicians: mean duration of connections | through study completion, an average of 11 months
Feasibility of the intervention for patients | through study completion, an average of 11 months
  number of screening failure and prematurely withdrawal
Feasibility of the intervention for technicians | through study completion, an average of 11 months
  duration of intervention
Feasibility of the intervention for nurses | through study completion, an average of 11 months
  response time following a notification
Technological performance indices of the system: failures in data transmission | through study completion, an average of 11 months
Technological performance indices of the system: inaccessibility | through study completion, an average of 11 months
Technological performance indices of the system: devices deficiencies | through study completion, an average of 11 months
  technical problems with any medical devices (leading or not to replacement).
Number of tele-notification per patient | through study completion, an average of 11 months
Frequency of tele-notifications per patient | through study completion, an average of 11 months
Patient care plan: number of changes implemented by investigators. | through study completion, an average of 11 months
Clinical events including medical consultations, hospitalizations and adverse events | through study completion, an average of 11 months
  Overall description of medical consultations, hospitalizations and adverse events. For adverse events, in addition, evaluation of seriousness and causal relationship with the medical device of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane SH Hominal, doctor, Principal Investigator — Centre hospitalier d'Annecy Genevois
Locations (6):
- France (6):
  - Cabinet Privé de Cardiologie - 2, rue jean jaurès, Annecy
  - Cabinet Privé de Pneumologie - 7 rue gabriel de mortillet, Annecy
  - Centre Hospitalier d'Annecy Genevois - service cardiologie - 1 avenue de l'Hôpital BP 90074 Metz-Tessy, Pringy
  - Centre Hospitalier d'Annecy Genevois - service pneumologie - 1 avenue de l'Hôpital BP 90074 Metz-Tessy, Pringy
  - Cabinet privé de pneumologie - 28 avenue de Genève, Saint-Julien-en-Genevois
  - cabinet privé de médecine générale - 18, rue Louis Haase, Thônes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkinson TM, Donaldson GC, Hurst JR, Seemungal TA, Wedzicha JA. Early therapy improves outcomes of exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1298-303. doi: 10.1164/rccm.200310-1443OC. Epub 2004 Feb 27. PMID 14990395
- [Background] Conway G. Case management for heart failure in the emergency department. Crit Pathw Cardiol. 2006 Mar;5(1):25-8. doi: 10.1097/01.hpc.0000202240.99184.81. PMID 18340214
- [Background] Elbert NJ, van Os-Medendorp H, van Renselaar W, Ekeland AG, Hakkaart-van Roijen L, Raat H, Nijsten TE, Pasmans SG. Effectiveness and cost-effectiveness of ehealth interventions in somatic diseases: a systematic review of systematic reviews and meta-analyses. J Med Internet Res. 2014 Apr 16;16(4):e110. doi: 10.2196/jmir.2790. PMID 24739471
- [Background] Marcolino MS, Maia JX, Alkmim MB, Boersma E, Ribeiro AL. Telemedicine application in the care of diabetes patients: systematic review and meta-analysis. PLoS One. 2013 Nov 8;8(11):e79246. doi: 10.1371/journal.pone.0079246. eCollection 2013. PMID 24250826
- [Background] Lundell S, Holmner A, Rehn B, Nyberg A, Wadell K. Telehealthcare in COPD: a systematic review and meta-analysis on physical outcomes and dyspnea. Respir Med. 2015 Jan;109(1):11-26. doi: 10.1016/j.rmed.2014.10.008. Epub 2014 Oct 27. PMID 25464906
- [Background] Cruz J, Brooks D, Marques A. Home telemonitoring effectiveness in COPD: a systematic review. Int J Clin Pract. 2014 Mar;68(3):369-78. doi: 10.1111/ijcp.12345. Epub 2014 Jan 28. PMID 24472009
- [Background] Goldstein RS, O'Hoski S. Telemedicine in COPD: time to pause. Chest. 2014 May;145(5):945-949. doi: 10.1378/chest.13-1656. PMID 24798834
- [Background] Conway A, Inglis SC, Chang AM, Horton-Breshears M, Cleland JG, Clark RA. Not all systematic reviews are systematic: a meta-review of the quality of systematic reviews for non-invasive remote monitoring in heart failure. J Telemed Telecare. 2013 Sep;19(6):326-37. doi: 10.1177/1357633X13503427. Epub 2013 Sep 25. PMID 24163297
- [Background] Nakamura N, Koga T, Iseki H. A meta-analysis of remote patient monitoring for chronic heart failure patients. J Telemed Telecare. 2014 Jan;20(1):11-7. doi: 10.1177/1357633X13517352. Epub 2013 Dec 18. PMID 24352899
- [Background] Purcell R, McInnes S, Halcomb EJ. Telemonitoring can assist in managing cardiovascular disease in primary care: a systematic review of systematic reviews. BMC Fam Pract. 2014 Mar 7;15:43. doi: 10.1186/1471-2296-15-43. PMID 24606887
- [Background] Kitsiou S, Pare G, Jaana M. Effects of home telemonitoring interventions on patients with chronic heart failure: an overview of systematic reviews. J Med Internet Res. 2015 Mar 12;17(3):e63. doi: 10.2196/jmir.4174. PMID 25768664
- [Background] Kotb A, Cameron C, Hsieh S, Wells G. Comparative effectiveness of different forms of telemedicine for individuals with heart failure (HF): a systematic review and network meta-analysis. PLoS One. 2015 Feb 25;10(2):e0118681. doi: 10.1371/journal.pone.0118681. eCollection 2015. PMID 25714962
- [Background] Pandor A, Gomersall T, Stevens JW, Wang J, Al-Mohammad A, Bakhai A, Cleland JG, Cowie MR, Wong R. Remote monitoring after recent hospital discharge in patients with heart failure: a systematic review and network meta-analysis. Heart. 2013 Dec;99(23):1717-26. doi: 10.1136/heartjnl-2013-303811. Epub 2013 May 16. PMID 23680885
- [Background] Feltner C, Jones CD, Cene CW, Zheng ZJ, Sueta CA, Coker-Schwimmer EJ, Arvanitis M, Lohr KN, Middleton JC, Jonas DE. Transitional care interventions to prevent readmissions for persons with heart failure: a systematic review and meta-analysis. Ann Intern Med. 2014 Jun 3;160(11):774-84. doi: 10.7326/M14-0083. PMID 24862840
- [Background] Kitsiou S, Pare G, Jaana M. Systematic reviews and meta-analyses of home telemonitoring interventions for patients with chronic diseases: a critical assessment of their methodological quality. J Med Internet Res. 2013 Jul 23;15(7):e150. doi: 10.2196/jmir.2770. PMID 23880072
- [Background] Ekeland AG, Bowes A, Flottorp S. Effectiveness of telemedicine: a systematic review of reviews. Int J Med Inform. 2010 Nov;79(11):736-71. doi: 10.1016/j.ijmedinf.2010.08.006. PMID 20884286
- [Background] Ekeland AG, Bowes A, Flottorp S. Methodologies for assessing telemedicine: a systematic review of reviews. Int J Med Inform. 2012 Jan;81(1):1-11. doi: 10.1016/j.ijmedinf.2011.10.009. Epub 2011 Nov 21. PMID 22104370
- [Background] Conway A, Inglis SC, Clark RA. Effective technologies for noninvasive remote monitoring in heart failure. Telemed J E Health. 2014 Jun;20(6):531-8. doi: 10.1089/tmj.2013.0267. Epub 2014 Apr 14. PMID 24731212
- [Background] Barnett K, Mercer SW, Norbury M, Watt G, Wyke S, Guthrie B. Epidemiology of multimorbidity and implications for health care, research, and medical education: a cross-sectional study. Lancet. 2012 Jul 7;380(9836):37-43. doi: 10.1016/S0140-6736(12)60240-2. Epub 2012 May 10. PMID 22579043
- [Background] Lefevre T, d'Ivernois JF, De Andrade V, Crozet C, Lombrail P, Gagnayre R. What do we mean by multimorbidity? An analysis of the literature on multimorbidity measures, associated factors, and impact on health services organization. Rev Epidemiol Sante Publique. 2014 Oct;62(5):305-14. doi: 10.1016/j.respe.2014.09.002. Epub 2014 Oct 25. PMID 25444838
- [Background] Smith SM, Soubhi H, Fortin M, Hudon C, O'Dowd T. Managing patients with multimorbidity: systematic review of interventions in primary care and community settings. BMJ. 2012 Sep 3;345:e5205. doi: 10.1136/bmj.e5205. PMID 22945950
- [Background] Fabbri LM, Boyd C, Boschetto P, Rabe KF, Buist AS, Yawn B, Leff B, Kent DM, Schunemann HJ; ATS/ERS Ad Hoc Committee on Integrating and Coordinating Efforts in COPD Guideline Development. How to integrate multiple comorbidities in guideline development: article 10 in Integrating and coordinating efforts in COPD guideline development. An official ATS/ERS workshop report. Proc Am Thorac Soc. 2012 Dec;9(5):274-81. doi: 10.1513/pats.201208-063ST. PMID 23256171
- [Background] Onder G, Palmer K, Navickas R, Jureviciene E, Mammarella F, Strandzheva M, Mannucci P, Pecorelli S, Marengoni A; Joint Action on Chronic Diseases and Promoting Healthy Ageing across the Life Cycle (JA-CHRODIS). Time to face the challenge of multimorbidity. A European perspective from the joint action on chronic diseases and promoting healthy ageing across the life cycle (JA-CHRODIS). Eur J Intern Med. 2015 Apr;26(3):157-9. doi: 10.1016/j.ejim.2015.02.020. Epub 2015 Mar 18. PMID 25797840
- [Background] Martin-Lesende I, Orruno E, Bilbao A, Vergara I, Cairo MC, Bayon JC, Reviriego E, Romo MI, Larranaga J, Asua J, Abad R, Recalde E. Impact of telemonitoring home care patients with heart failure or chronic lung disease from primary care on healthcare resource use (the TELBIL study randomised controlled trial). BMC Health Serv Res. 2013 Mar 28;13:118. doi: 10.1186/1472-6963-13-118. PMID 23537332
- [Background] Sutherland D, Hayter M. Structured review: evaluating the effectiveness of nurse case managers in improving health outcomes in three major chronic diseases. J Clin Nurs. 2009 Nov;18(21):2978-92. doi: 10.1111/j.1365-2702.2009.02900.x. Epub 2009 Sep 11. PMID 19747197
- [Background] Chow SK, Wong FK. A randomized controlled trial of a nurse-led case management programme for hospital-discharged older adults with co-morbidities. J Adv Nurs. 2014 Oct;70(10):2257-71. doi: 10.1111/jan.12375. Epub 2014 Mar 12. PMID 24617755
- [Background] Prochaska JO, DiClemente CC. Transtheorical therapy toward a more integrative model of change. Psychotherapy: Theory, Research and Practice, 1982;19(3):276-287
- [Result] Chacornac M, Faoro A, Texereau J, Billoet C, Hominal S. Performance of an eHealth (NOMHAD) System Comprising Telemonitoring, Telenotification, and Telecoaching for Patients With Multimorbidity: Proof-of-Concept Study. JMIR Form Res. 2022 Mar 11;6(3):e32205. doi: 10.2196/32205. PMID 35275068